CLINICAL TRIAL: NCT02389010
Title: Clinical Efficacy of Platelet Gel From Cord Blood for the Treatment of Diabetic Foot Ulcers
Acronym: CBPG-DFU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Nazionale Sangue (Other Government)
Collaborators: Italian National Cord Blood Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-02

CONDITIONS: Diabetic Foot Ulcers
Keywords: Umbilical Cord Blood; Diabetic Foot; Ulcer; Cost; Effectiveness; Safety; Platelet Gel; Cord Blood Platelet Gel; Adverse Event
MeSH Terms: conditions — Diabetic Foot; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allogeneic Cord Blood Platelet Gel-CBPG (Experimental): For the medication of patients, one CBPG unit (mean volume 10 mL, range 5-15; mean platelet concentration 1 x 109/L, range 0.8 - 1.2 x 109/L. 10 mL in plasma) will be administered every 3-4 days. CBPG units, cryopreserved and stored in a plastic bag in a -80°C freezer, will be thawed at 37°C in a waterbath and activated with Calcium gluconate and immediately transported to sites of clinical use and applied to the skin ulcer without breaking the sterility chain.
  Interventions: Biological: Allogeneic cord blood platelet gel-CBPG
- Standard Local Medications-SLM (Active Comparator): 1 administration every 3-4 days for 4 weeks. Each clinical center will use their validated standard local medications. Details and specifications of the local standard medication procedures will be collected from each participating centre.
  Interventions: Other: Standard Local Medications-SLM

INTERVENTIONS:
Biological: Allogeneic cord blood platelet gel-CBPG — For the medication of patients, one CBPG unit (mean volume 10 mL, range 5-15; mean platelet concentration 1 x 109/L, range 0.8 - 1.2 x 109/L. 10 mL in plasma) will be administered every 3-4 days. CBPG units, cryopreserved and stored in a plastic bag in a -80°C freezer, will be thawed at 37°C in a waterbath and activated with Calcium gluconate and immediately transported to sites of clinical use and applied to the skin ulcer without breaking the sterility chain.
  Arms: Allogeneic Cord Blood Platelet Gel-CBPG
Other: Standard Local Medications-SLM — Each clinical center will use their validated standard local medications. Details and specifications of the local standard medication procedures will be collected from each participating centre.
  Arms: Standard Local Medications-SLM

SUMMARY:
A novel method (PCT n. WO 2010/007502 A2, 2010) has been developed to obtain platelet gel from umbilical cord blood (CBPG). The main advantages so far identified in CBPG as compared to platelet gel derived from adult platelets relate to the lack of microbiological contamination in the former and to a different profile of growth factors concentrations, such as a higher content of VEGF and lower content of TGF in CBPG. Recent developments have led to a procedure in which CBPG can be prepared, stored in a cryopreservation bag and applied to the skin ulcer without breaking the sterility chain. In spite of promising results on allogeneic CBPG, a randomized clinical trial of sufficient statistical power to detect significant advantages (clinical and economical) will be performed in patients affected by diabetic foot ulcers and randomly treated with CBPG versus standard local medications (SLM).This study is a multicenter (8 centers) controlled randomized clinical trial. Outcomes: (1) primary objective is to evaluate the number of closed skin ulcers within 4 weeks of treatment with CBPG vs standard local medications; (2) secondary objectives are percent skin ulcer closure area, number and type of adverse events and cost of treatment. Sample size calculation: 95 + 5 (dropout) test and 95 + 5 (dropout) control patients ensure 80% power to detect as statistically significant (p<0.05) >60% healing in test vs 40% healing in control.Each clinical centre has been invited to enrol 15 treated and 15 control patients, according to local availability in 12 months. CB units are routinely collected after mother's informed consent before and after placenta delivery in accredited public cord blood banks belonging to the Italian Cord Blood Network (ITCBN) coordinated by the Centro Nazionale Sangue (CNS). After storage and transportation at monitored room temperature, the units will be processed for the preparation of CBPG within 48 hours of collection. CBPG will be prepared according to standard procedures with a defined final platelet concentration (0.8-1.2 x 109/L). The CBPC units will be finally cryopreserved in a -80°C freezer in view of the clinical use of the CBPG, which will require thawing at 37°C in a waterbath and activation with Calcium gluconate. For SLM, each clinical center will use their validated standard procedures.

DETAILED DESCRIPTION:
Background information and study rationale: Evidence no. 1 (platelet gel). The gel obtained upon platelet activation of platelet rich plasma with thrombin or with pharmaceutical extracts of cobra venom is a blood component that has been used for clinical purposes for a number of years. The rationale supporting this therapy relates to the high content of growth factors in platelet alpha granules that can be delivered topically by a natural biocompatible carrier (i.e. the platelets) upon platelet activation. So far, platelet gel has been mainly used to repair recalcitrant skin ulcers in diabetic and non-diabetic patients in an autologous blood donation setting. Unfortunately, most candidates to this therapy are elderly patients, frequently affected by a number of pathologic conditions and comorbidities which make them mostly unfit or unsuitable for the process of autologous blood collection. In practice, most patients who could mostly benefit from this therapy are de facto deprived of a potentially effective treatment because of this limitation.

Evidence no. 2 (blood transfusion safety). Current systems for blood donor screening by viral nucleic acid testing have dramatically reduced the risk of transmission of infectious conditions through the transfusion of blood and blood components. Accordingly, limitations to the use of allogeneic blood and blood components that were mandatory some decades ago do not find current justification. This opens the perspective of an increased use of allogeneic blood components - including platelet gel - with potential advantages for large numbers of patients in whom they are mostly indicated.

Evidence no. 3 (platelet gel from cord blood). A research group led by the investigator proposing the present project has recently developed a novel method (PCT no. WO 2010/007502 A2, 21 January 2010) to obtain platelet gel from the newborn's blood remaining in the placenta after delivery, aka umbilical cord blood or placental blood. The main advantages so far identified in platelet gel derived from cord blood platelets as compared to platelet gel derived from adult platelets relate to the lack of microbiological contamination in the former and to a different profile of growth factors concentrations, the main difference consisting in a higher content of VEGF and lower content of TGF in cord blood platelet gel. Recent modifications performed have led to a procedure in which platelet gel from cord blood can be prepared and stored in a small plastic bag rather than in tubes or dishes, which can be easily cryopreserved, stored, transported to sites of clinical use and applied to the skin ulcer without breaking the sterility chain. This paves the way for a broader use of allogeneic cord blood platelet gel inside and outside hospitals.

Evidence no. 4 (knowledge gaps). In spite of interesting and promising results on allogeneic cord blood platelet gel, three elements are missing before the latter may be used extensively in patients who may need it: (1) a more complete biochemical characterization; (2) a regional or national program to collect and prepare the necessary doses of cord blood platelet gel; (3) a randomized clinical trial of sufficient statistical power to detect significant advantages (both clinical and economical) in patients treated with cord blood platelet gel versus controls treated with skin ulcer advanced medications. In this regard, small scale investigations suggest that the effective use of platelet gel may reduce recalcitrant skin ulcer medication costs to one tenth of costs currently reimbursed to hospitals for ineffective advanced medication (from about 190.000 euro to about 19.000 euro to treat 11 elderly patients).

Evidence no. 5 (cord blood banking and transplant). Cord blood - which was once disposed as a hospital waste - is currently a precious source of hemopoietic stem cells to be used for bone marrow replacement in patients affected by severe blood diseases. The last 25 years of clinical experience with this stem cell source has shown that high cell dose and better HLA match are the most important factors impacting on patient survival. For this reason, cord blood banks preferentially cryopreserve cord blood units with very large volumes, as volume correlates with cell content, and discard about three quarters of units collected. It is expected that the discard rate will increase in the future, also because the worldwide inventory of about 600.000 cord blood units in 128 cord blood banks already includes units with volumes that are currently considered sub-optimal for hemopoietic transplant. It is therefore expected that 70-80% of cord blood units donated for allogeneic hemopoietic transplant may be unsuitable for this use and ultimately discarded. These units can be used for the preparation of platelet gel if a suitable program of recovery from delivery suites, transportation to a production site and processing into platelet gel is developed.

Study design: This study is a multicenter controlled randomized clinical trial (Allogeneic cord blood platelet gel (CBPG) vs Standard local medications (SLM)). Each clinical centre has been invited to enroll 15 treated and 15 control patients, according to local availability in the 12 month study interval.

Sample size calculation : 95 + 5 (dropout) test and 95 + 5 (dropout) control patients ensure 80% power to detect as statistically significant (p<0.05) >60% healing in test vs 40% healing in controls (Pocock, 1983).

Principles of Statistical analysis: Descriptive statistics: summary tables by treatment group (except for baseline characteristics which will be provided by sequence and overall) according to the type of variable summarised; quantitative criteria: standard quantitative statistics (N, mean, SD, median, min-max); qualitative criteria: frequency distribution [number of non-missing observations (N) and percentages (%)].

CBPG preparation and quality control: CB units are routinely collected after mother's informed consent in plastic bags containing 21-29 mL of citrate-phosphate-dextrose (CPD) anticoagulant by trained midwives, before and after placenta delivery in natural deliveries and in cesarean sections respectively, according to locally validated standard operation procedures, in accredited public cord blood banks belonging to the Italian Cord Blood Network coordinated by the Centro Nazionale Sangue. After storage and transportation at monitored room temperature, the units will be processed for the preparation of CBPG within 48 hours of collection. Based on a previous standardization exercise, the participating banks will be allowed to use locally available bags of convenient size and nominal volume that they consider appropriate for this protocol. In the above standardization exercise, it was decided to define the main characteristics of the final CBPC as follows: target mean volume 10 ml, range 5-15; target mean platelet concentration 1 x 109/L, range 0.8 - 1.2 x 109/L. The latter concentration was selected in agreement with the platelet concentration defined by the Italian Society of Transfusion Medicine for platelet gel obtained from adult blood. CBPG will be prepared according to procedures defined during pilot studies at each bank, which included an initial centrifugation of CB at 200-210 g x 10-15 minutes, followed by the transfer of the platelet rich plasma (PRP) into a secondary bag, centrifugation of the PRP at 1800-2600 g x 15 minutes and removal of the supernatant platelet poor plasma (PPP) in excess of the final target volume of the CBPC. The latter was defined by an automated algorithm performed by an Excel spreadsheet used for data collection, which takes into account the platelet concentration in the PRP and the minimum (0.8 x 109/L) and maximum (1.2 x 109/L) values of the platelet concentration aimed at in the final CBPC. The platelet concentrations in the PRP divided by 0.8 and by 1.2 x 109/L provide the upper and lower bounds of the CBPC volume respectively. The final volume was set by determining the net weight of the CBPC on an electronic scale. The CBPC units will be finally cryopreserved in a -80 °C mechanical freezer in view of the clinical use of the CBPG, which will require thawing at 37° C in a waterbath and activation with Calcium gluconate. For the standard local medications, each clinical center will use their validated standard local medications. Details and specifications of the local standard medication procedures will be collected from each participating centre.

Treatments: Test treatments: CBPG is a gel formed by fibrin trapping platelet fragments from about 10 billion platelets in 10 mL of neonatal plasma anticoagulated with CPD. It is stored in a commercial PVC bag for blood component preparation and storage.

In the '80s, David Knighton developed a technique for in vitro stimulation of platelets, with thrombin solutions that allowed to collect a supernatant abundant of growth factors. This product, derived from patient platelets was locally applied as gel to encourage the ulcer repair.

The rationale in the use of such product is in the presence of several tissue growth factors: P.D.G.F. (Platelet Derived Growth Factor); E.G.F. (Epidermal Growth Factor); T.G.F. (Transforming Growth Factor); V.E.G.F. (Vascular Endothelial Growth Factor); I.G.F. 1 e 2 (Insulin Growth Factor 1 and 2); F.G.F. (Fibroblast Growth Factor). Applying in situ the iper-concentrated and activated platelets as platelet gel, tissue regeneration processes are started and accelerated. In this setting, platelets are similar to cellular laboratory-tanks that process, store and then release (if activated) several growth factors able to stimulate mesenchymal stem cell regeneration as fibroblasts, osteoblasts and endothelial cells. This platelet ability to take part in tissue repair mechanisms has been the theoretical essential requirement to use the platelet gel in several circumstances, all associated with the requirement of tissue repair activation.

Repeated PG applications have been shown to be useful prior to wound surgery since they can reduce lesion size, improve anatomic and morphological conditions of wound bed and margins and trigger neo-angiogenesis at the margins and within the necrotic area.

Usual source of platelet fractions is adult human blood, but this source involves relevant drawbacks and problems. Peripheral blood from a human cannot be used without potential risks due to alloreactivity, resulting in several clinical complications. On the other hand, the availability of autologous blood is generally low, since it can be dangerous to withdraw a sufficient amount from a patient who cannot tolerate such a withdrawal. Moreover, allogeneic blood from adult donors can involve risks of infections.

Platelet fractions derived from human placental blood can avoid the above drawbacks and also contain high concentrations of platelet factors.

Dosage and Administration: For the medication of patients enrolled in the treatment arm, one CBPG unit (mean volume 10 ml, range 5-15; mean platelet concentration 1 x 109/L (0.8 - 1.2 x 109/L) will be administered every 3-4 days. CBPG units, cryopreserved and stored in a small plastic bag in a -80°C freezer, will be thawed at 37°C in a waterbath and activated with Calcium gluconate and immediately transported to sites of clinical use and applied to the skin ulcer without breaking the sterility chain.

Efficacy assessment: Efficacy will be evaluated with the CBPG-DFU Clinical Research Form.

Safety assessments: Information will be collected on all adverse events and on events associated with CBPG that will occur during treatment. Care and management efforts provided at each treatment visit will include cleansing and assessing the wound and obtaining vital signs and an interim wound history, including information regarding adverse events, concomitant medications, nutrition and weight-bearing status.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years
2. Patient with diabetic foot ulcers
3. Size of ulcer (5 cm^2 < X < 30 cm^2)
4. Absence of undermining or tunneling
5. TUC I and II C. At the time of 1st application, ulcer is not clinically infected (smelly, perilesional edematous tissue, hot and flushed)
6. Effective Revascularization ( TcPO2 foot >30 mmHg and Patency of one or more tibial arteries until the ankle/foot)
7. Informed consent
8. Patient able to understand the conditions of the study and to participate for its entire duration

Exclusion criteria

1. Patient with serious medical conditions that contraindicate the patient's participation in the study
2. Ineffective revascularization
3. Heel ulcer and outcomes of amputation
4. Patient with present clinical infection
5. Bone and/or sinew exposure
6. Current pregnancy
7. Use of experimental drugs.
8. Negative Pressure (possible use in control arm patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of closed skin ulcers within 4 weeks of treatment with cord blood platelet gel (CBPG) vs standard local medications | 4 weeks
  The major end-point will be to test feasibility and compare efficacy of treating diabetic foot skin ulcers (Texas C I-II) with allogeneic CBPG versus SLM and their respective costs. The primary outcome measures will be: number of healed wounds after 4 weeks of CBPG treatment versus control and time to achieve complete closure. Lesions will be assessed two times per week. Wounds with less than 50% closure after 4 weeks will be considered as a failure. The main target will be to validate the clinical use of an allogeneic product matching several requirements: to comply with routine process of periodic blood collection and blood component preparation; to maintain closed and aseptic conditions through the entire process; to contain platelet growth factor concentrations reported to be clinically effective; to be suitable to treat one medium-size ulcer per aliquot, defined as 'CBPG unit' (on average 10 mL of CB plasma containing 10 billion platelets); to be ABO compatible with the patient.

SECONDARY OUTCOMES:
Percent skin ulcer closure area | 4 weeks
Number and type of adverse events | 4 weeks
Cost of treatment | 4 weeks
  Cost analysis will include costs associated with blood component preparation, storage and activation; the administration of CBPG or standard local medications; dressing materials; and personnel workload (technicians and nurses).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Marconi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Simonetta Pupella, MD, Study Chair — Centro Nazionale Sangue
Locations (9):
- Italy (8):
  - Ospedaliero-Universitaria di Bologna, Bologna
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Presidio Ospedaliero "Spirito Santo", Pescara
  - Azienda Ospedalero-Universitaria Pisana, Pisa
  - Presidio Ospedaliero "E. Morelli", Reggio Calabria
  - Policlinico Umberto I - "Sapienza" Università di Roma, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- Hospital de la Santa Creu i Sant Pau - Servicio de Angiología, Cirugía Vascular y Endovascular, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosso L, Parazzi V, Damarco F, Righi I, Santambrogio L, Rebulla P, Gatti S, Ferrero S, Nosotti M, Lazzari L. Pleural tissue repair with cord blood platelet gel. Blood Transfus. 2014 Jan;12 Suppl 1(Suppl 1):s235-42. doi: 10.2450/2013.0214-12. Epub 2013 May 14. PMID 23736928
- [Result] Parazzi V, Lazzari L, Rebulla P. Platelet gel from cord blood: a novel tool for tissue engineering. Platelets. 2010;21(7):549-54. doi: 10.3109/09537104.2010.514626. PMID 20873963
- [Result] Giusti I, Rughetti A, D'Ascenzo S, Millimaggi D, Pavan A, Dell'Orso L, Dolo V. Identification of an optimal concentration of platelet gel for promoting angiogenesis in human endothelial cells. Transfusion. 2009 Apr;49(4):771-8. doi: 10.1111/j.1537-2995.2008.02033.x. Epub 2008 Dec 23. PMID 19170984
- [Result] Mishra A, Woodall J Jr, Vieira A. Treatment of tendon and muscle using platelet-rich plasma. Clin Sports Med. 2009 Jan;28(1):113-25. doi: 10.1016/j.csm.2008.08.007. PMID 19064169
- [Result] Spyridakis M, Christodoulidis G, Chatzitheofilou C, Symeonidis D, Tepetes K. The role of the platelet-rich plasma in accelerating the wound-healing process and recovery in patients being operated for pilonidal sinus disease: preliminary results. World J Surg. 2009 Aug;33(8):1764-9. doi: 10.1007/s00268-009-0046-y. PMID 19424751
- [Result] O'Connell SM, Impeduglia T, Hessler K, Wang XJ, Carroll RJ, Dardik H. Autologous platelet-rich fibrin matrix as cell therapy in the healing of chronic lower-extremity ulcers. Wound Repair Regen. 2008 Nov-Dec;16(6):749-56. doi: 10.1111/j.1524-475X.2008.00426.x. PMID 19128245
- [Result] Gope ML, Gope R. Tyrosine phosphorylation of EGF-R and PDGF-R proteins during acute cutaneous wound healing process in mice. Wound Repair Regen. 2009 Jan-Feb;17(1):71-9. doi: 10.1111/j.1524-475X.2008.00443.x. PMID 19152653
- [Result] Nikolidakis D, Jansen JA. The biology of platelet-rich plasma and its application in oral surgery: literature review. Tissue Eng Part B Rev. 2008 Sep;14(3):249-58. doi: 10.1089/ten.teb.2008.0062. PMID 18601587
- [Result] Knighton DR, Ciresi KF, Fiegel VD, Austin LL, Butler EL. Classification and treatment of chronic nonhealing wounds. Successful treatment with autologous platelet-derived wound healing factors (PDWHF). Ann Surg. 1986 Sep;204(3):322-30. doi: 10.1097/00000658-198609000-00011. PMID 3753059
- [Result] Knighton DR, Ciresi K, Fiegel VD, Schumerth S, Butler E, Cerra F. Stimulation of repair in chronic, nonhealing, cutaneous ulcers using platelet-derived wound healing formula. Surg Gynecol Obstet. 1990 Jan;170(1):56-60. PMID 2403699
- See also: Competent authority website — http://www.centronazionalesangue.it